CLINICAL TRIAL: NCT03666026
Title: Improving Influenza Vaccination Delivery Across a Health System by the Electronic Health Records Patient Portal
Brief Title: Patient Portal - Flu Reminder Recall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Clinical Research, UCLA David Geffen School of Medicine, Dept of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889; 1R01AI135029-01 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Influenza; Respiratory Tract Infections; Vaccines
Keywords: Reminder Recall (R/R); Influenza Vaccine; Electronic Health Record
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care control (No Intervention): Participants in this group will not receive any MyChart influenza vaccination reminders
- 1 MyChart R/R (Experimental): Participants in this group will receive up to 1 influenza reminder recall notice via their MyChart account
  Interventions: Behavioral: 1 MyChart R/R
- 2 MyChart R/R (Experimental): Participants in this group will receive up to 2 influenza reminder recall notices via their MyChart account
  Interventions: Behavioral: 2 MyChart R/R
- 3 MyChart R/R (Experimental): Participants in this group will receive up to 3 influenza reminder recall notices via their MyChart account
  Interventions: Behavioral: 3 MyChart R/R

INTERVENTIONS:
Behavioral: 1 MyChart R/R — Up to 1 flu vaccine reminder recall notice sent via MyChart to patients who are due for the flu vaccine, per the EMR records of the health system.
  Arms: 1 MyChart R/R
Behavioral: 2 MyChart R/R — Up to 2 flu vaccine reminder recall notices sent every 3-4 weeks via MyChart to patients who are due for the flu vaccine, per the EMR records of the health system.
  Arms: 2 MyChart R/R
Behavioral: 3 MyChart R/R — Up to 3 flu vaccine reminder recall notices sent every 3-4 weeks via MyChart to patients who are due for the flu vaccine, per the EMR records of the health system.
  Arms: 3 MyChart R/R

SUMMARY:
This trial is taking place in Los Angeles, CA at clinics within the UCLA Health System.

Despite the Advisory Committee on Immunization Practices (ACIP) recommendation in 2010 that all people above 6 months of age should receive an annual flu vaccine, vaccination rates remain low: at 6m-4.9 yrs. (70%), 5-17.9 yrs. (56%), 18-64.9 yrs. (38%), and >65 yrs. (63%). The investigators will assess the effectiveness and cost-effectiveness of 1, 2, 3 MyChart R/R messages as compared to the standard of care control (no messages).

DETAILED DESCRIPTION:
Annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs. Concerns about pandemic influenza elevate the need to prevent flu outbreaks.

Numerous studies, including Cochrane or systematic reviews, and reports by the CDC and the Task Force on Community Preventive Services, highlight 4 evidence-based strategies to raise child and adult influenza vaccination rates: 1) increase patient demand by reminder-recall or education, 2) expand patient access to influenza vaccinations (e.g., flu vaccine clinics), 3) implement provider strategies such as prompts or standing orders, and 4) use societal strategies (e.g., reducing costs).

Reminder/recall (R/R), sent by phone, mail or other modality, can improve child and adult influenza vaccination rates. However, fewer than one-fifth of pediatric or adult primary care practices utilize patient R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients.

A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are used by about half of Americans and half of UCLA patients. Portals can theoretically improve upon phone, mail or text R/R by adding information such as web links, videos, or images, allowing patients to schedule their own visits, and linking to the medical chart to customize messages.

For this randomized control trial, the intent is to evaluate the impact of patient portal (MyChart) reminder recalls - either 1, 2, or 3 reminders versus the standard of care control group, specifically in relation to raising influenza vaccination rates among UCLA Health System's primary care patients aged 6 months and older.

The proposed design of this 4-arm RCT:

1. Standard of care control (no messages)
2. Up to 1 portal R/R messages
3. Up to 2 portal R/R messages
4. Up to 3 portal R/R messages

Hypothesis 1: >1 portal R/R will increase vaccination rates vs. no R/R. Hypothesis 2: More R/R messages will raise vaccination rates (3R/R > 2R/R > 1R/R > 0R/R).

For the primary analysis, only the data from the randomly selected index patients (1 index patient per household) will be included.

For relevant study arms, the first R/R message will be sent in October 2018.

ELIGIBILITY:
Inclusion Criteria:

• A patient within the UCLA Health System identified by the system as a primary care patient per an internal algorithm, with a documented primary care visit within the last 3 years as of 8/1/18.

Exclusion Criteria:

• A patient not identified by the UCLA Health System's internal algorithm as a primary care patient.

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164205 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be prepared for publication at the end of the trial.

REFERENCES:
- [Derived] Szilagyi PG, Albertin C, Casillas A, Valderrama R, Duru OK, Ong MK, Vangala S, Tseng CH, Rand CM, Humiston SG, Evans S, Sloyan M, Lerner C. Effect of Patient Portal Reminders Sent by a Health Care System on Influenza Vaccination Rates: A Randomized Clinical Trial. JAMA Intern Med. 2020 Jul 1;180(7):962-970. doi: 10.1001/jamainternmed.2020.1602. PMID 32421168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care Control | 1 MyChart R/R | 2 MyChart R/R | 3 MyChart R/R
Started | 41070 | 41055 | 41046 | 41034
Completed | 41070 | 41055 | 41046 | 41034
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were eligible for study participation if they were at least 6 months of age at the start of intervention (ie, eligible for influenza vaccination), a primary care patient within the UCLA Health System according to the health system's criteria, and an active patient portal user (≥1 log-in during the past 12 months), other than initial account log-in.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Control | 1 MyChart R/R | 2 MyChart R/R | 3 MyChart R/R | Total
Number analyzed (Participants) | 41070 | 41055 | 41046 | 41034 | 164205
Age, Customized [Number; unit: Percent of participants]
  0.5-17 years 0-5 years | 7.4 | 7.3 | 7.3 | 7.4 | 7.4
  18-64 years | 73.8 | 73.9 | 74.1 | 74.0 | 74.0
  >= 65 years | 18.8 | 18.8 | 18.6 | 18.5 | 18.7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23985 | 23935 | 23889 | 23964 | 95773
  Male | 17085 | 17120 | 17157 | 17070 | 68432
Race/Ethnicity, Customized [Number; unit: Percent of participants]
  White | 57.3 | 57.5 | 57.2 | 57.1 | 57.3
  Black | 4.4 | 4.6 | 4.7 | 4.8 | 4.6
  Asian | 10.1 | 10.4 | 10.3 | 10.3 | 10.3
  Unkown | 28.2 | 27.6 | 27.7 | 27.9 | 27.8
  Hispanic Ethnicity | 46.9 | 46.7 | 46.7 | 47.0 | 46.9
Received influenza vaccination in prior two years [Number; unit: Percent of participants] | 46.9 | 46.7 | 46.7 | 47.0 | 46.9

OUTCOME MEASURES:

1. Primary Outcome: 1.Receipt of the Annual Influenza Vaccine (Between 10/1/18 - 4/2/19) Among Index Patients. Outcomes Will be Assessed Via Vaccine Data Extraction From the Electronic Health Record and External Claims and Pharmacy Data.
Description: Number of participants in each arm who received influenza vaccination
Time Frame: October 1, 2018 to April 2, 2019 during influenza vaccination season
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Control | 1 MyChart R/R | 2 MyChart R/R | 3 MyChart R/R
Number analyzed (Participants) | 41070 | 41055 | 41046 | 41034
Participants | 15385 | 15604 | 15660 | 15673
Statistical Analysis 1: Comparison: Standard of Care Control vs 1 MyChart R/R; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.03]
Statistical Analysis 2: Comparison: Standard of Care Control vs 2 MyChart R/R; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.04]
Statistical Analysis 3: Comparison: Standard of Care Control vs 3 MyChart R/R; Test type: Superiority; Risk Ratio (RR) = 1.02, 95% CI 2-sided [1.00 to 1.04]

ADVERSE EVENTS:
Time Frame: This pragmatic, 4-arm randomized clinical trial was performed from October 1, 2018, to April 2, 2019, across the UCLA (University of California, Los Angeles) health care system. A total of 164 205 patients in 52 primary care practices who had used the patient portal within 12 months were included. Adverse events were not assessed/monitored.
Description: We conducted a trial of whether reminder sent via the portal impacted influenza vaccination rates; we did not collect adverse event or serious event information.
Arm/Group | Standard of Care Control | 1 MyChart R/R | 2 MyChart R/R | 3 MyChart R/R
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03666026/Prot_SAP_000.pdf